CLINICAL TRIAL: NCT02144038
Title: A Phase Ib/II, Multi-center, Study of Oral LGH447 in Combination With Oral BYL719 in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Study of the Safety and Effectiveness of LGH447 and BYL719 in Patients With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLGH447X2103C; 2013-004959-21 (EudraCT Number)
Record Dates: First submitted 2014-05-01; First posted 2014-05-21 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2018-04

CONDITIONS: Relapsed and Refractory Multiple Myeloma
Keywords: multiple myeloma,; relapsed and refractory,; LGH447,; pan-PIM inhibitor,; PIM Kinase,; BYL719,; PI3K inhibitor
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — LGH-447; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase Ib: LGH447 + BYL719 (Experimental): Dose-escalation, LGH447 in combinatinon with BYL719
  Interventions: Drug: LGH447; Drug: BYL719
- Phase II: LGH447 + BYL719 (Experimental): LGH447 + BYL719 (dosing according to MTD/RP2D from Phase Ib portion of the study)
  Interventions: Drug: LGH447; Drug: BYL719
- Phase II: LGH447 alone (Experimental): LGH447 alone (dosing according to single-agent RDE)
  Interventions: Drug: LGH447

INTERVENTIONS:
Drug: LGH447 — pan-PIM inhibitor
Drug: BYL719 — PI3K-alpha inhibitor
  Arms: Phase II: LGH447 + BYL719; Phase Ib: LGH447 + BYL719

SUMMARY:
This is a Phase Ib/II study with the primary purpose of the Phase Ib part being to estimate the MTD and/or recommended phase 2 dose (RP2D) of the combination of LGH447 and BYL719 when administered orally to adult patients with relapsed and refractory multiple myeloma. Once the MTD and/or RP2D is determined for the combination of LGH447 and BYL719, additional patients will be enrolled in the Phase II part to determine whether the combination of LGH447 and BYL719 exhibits improved anti-multiple myeloma activity compared to single agent LGH447. This trial never made it to the Phase II part of the this trial.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Patients with a confirmed diagnosis of multiple myeloma who have received two or more lines of therapy and are refractory to their most recent line of therapy, as defined as relapse while on therapy or within 60 days from their last line of therapy. If patient has not received either an immunomodulatory drug (IMID) or proteasome inhibitor as a prior therapy then Investigator must notify Novartis prior to the patient enrollment. Patients who have received a prior bone marrow transplant and otherwise meet the inclusion criteria are eligible for this study
* For patients in the Phase II portion of the study, must have measurable disease defined by at least 1 of the following 3 measurements:

  * Serum M-protein ≥ 0.5 g/dL
  * Urine M-protein ≥ 200 mg/24 hours OR
  * Serum free light chain (FLC) > 100 mg/L of involved FLC
* All patients must be willing to undergo a mandatory bone marrow aspirate and/or biopsy at baseline for the assessment of biomarker/pharmacodynamics and disease status

Exclusion Criteria:

* Systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any experimental therapy within 14 days or 5 half-lives, whichever is shorter, before the first dose of either study drug
* Radiotherapy within 14 days before the first dose of either study drug except localized radiation therapy for lytic bone lesions and plasmacytomas
* Major surgery within 2 weeks before the first dose of either study drug
* Ongoing therapy with chronic or high dose corticosteroids. Low dose steroids (i.e. prednisone ≤ 10 mg or an equivalent steroid dose), inhaled and topical steroids are permitted
* Patients who are currently receiving treatment with a prohibited medication that cannot be discontinued at least one week prior to the start of treatment:
* Narrow Therapeutic index substrates, strong inhibitors and strong inducers of CYP3A4
* Strong Inhibitors of CYP2D6
* Narrow therapeutic index substrates of CYP2C8, CYP2C9, CYP2C19 and CYP2D6
* Any of the following clinical laboratory results during screening (i.e., within 28 days before the first dose of either study drug):
* Absolute neutrophil count (ANC) < 1,000/mm3 without growth factor support within 7 days prior to testing
* Platelet count < 75,000 mm3 without transfusion support within 7 days prior to testing
* Bilirubin > 1.5 times the upper limit of the normal range (ULN).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the ULN.
* Calculated creatinine clearance < 30 ml/min according to Cockcroft-Gault equation
* Corrected QT interval (QTc) of > 450 milliseconds (ms) in males and > 470 milliseconds (ms) in females on baseline electrocardiogram (ECG) (using Fridericia [QTcF] corrected QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2015-10-28 (Actual); Study Completion 2015-10-28 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Number of Total Dose-limiting Toxicities (DLT) | Cycle 1 (28 days)
  Using a Bayesian logistic regression model (BLRM) to guide dose escalation and predict MTD or determine the RP2D for LGH447 in combination with BYL719 in relapsed and refractory multiple myeloma. The frequency and characteristics of DLTs will be assessed.
Phase II: Overall Response Rate (ORR) as assessed by Investigators | 29 months (End of Study)
  The proportion of patients with a confirmed best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) as assessed by Investigators using the International Myeloma Working group (IMWG) Criteria with modifications.
  End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.

SECONDARY OUTCOMES:
Phase II: Percent change of ORR (Overall Response Rate) between the two arms | 29 months (End of Study)
  The ORR percent change between the two arms, LGH447 in combination with BYL719 and LGH447 alone, is the parameter of interest. Both observed and Bayesian estimates of ORR percent change along with 80% confidence intervals and credible intervals will be calculated. End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.
Number of participants with adverse events, serious adverse events, changes in laboratory values, and electrocardiograms (ECGs), as a measure of safety and tolerability. | 23 months
  Assessments consisted of recording all adverse events (AEs) and serious adverse events (SAEs), the regular monitoring of hematology, blood chemistry, urinalysis, and coagulation parameters, as well as electrocardiograms.
Determine single and multiple dose Pharmacokinetics (PK) profiles | Approximately 8 months
  To determine the single and multiple dose PK profiles of the LGH447 and BYL719 combination (Phase Ib and II) and LGH447 alone (Phase II), by measuring plasma concentrations of LGH447 and BYL719 respectively at different timepoints prior and post study drug combination dosing on several days within cycle 1 and subsequent cycles for all patients in the Phase 1b and for the first 15 patients in each arm in the Phase 2 portion of the study. PK parameters including but not limited to Cmax, AUCinf, AUClast, AUCtau,T1/2, Tmax, Racc, CL/F, and Vz/F
Changes between pre- and post-treatment levels of pS6RP and 4EBP1 levels in bone marrow aspirates and 4EBP1 in peripheral blood | baseline, Cycle 2 Day 1
  Cycle 2 = 28 days; LGH447-mediated target modulation of the PIM pathway will be assessed from the collection of bone marrow biopsy and/or aspirates by flow cytometry, immunohistochemistry, or other methods as deemed appropriate. Decreases in the phosphorylation of markers (eg. S6RP and 4EBP1) will be measured in both pre- and post-dose bone marrow aspirate samples and peripheral blood samples.
Phase II: Absolute difference in ORR | 29 months (End of Study)
  Both observed and Bayesian estimates of absolute difference in ORR between the two arms will be calculated. The 80% confidence intervals and credible intervals for the difference will be provided. End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.
Disease Control Rate | 29 months (End of Study)
  Proportion of patients with a best overall response of sCR, CR, VGPR, PR, MR, or SD, using International Myeloma Working Group Criteria with modification. End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.
Progression Free Survival | 29 months (End of Study)
  Defined as the time from start of treatment to the date of event defined as the first documented PD/relapse, or death due to any cause, whichever comes first. End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.
Time to response | 29 months (End of Study)
  The time between date of randomization until first documented best overall response (sCR, CR, VPGR or PR). End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.
Duration of Response | 29 months (End of Study)
  Defined as the duration from the first documented onset of PR or better response to the date of documented PD/relapse or death due to multiple myeloma. End of Study (defined as the time when all patients have completed at least 6 cycles of treatment or discontinued treatment, or have been lost to follow up, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (3):
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(SC), Houston, Texas
  - Seattle Cancer Care Alliance Oncology Dept, Seattle, Washington
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Dept of Onc., Madison, Wisconsin
- Novartis Investigative Site, Prahran, Victoria, Australia
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Singapore, Singapore

REFERENCES:
- See also: Results for CLGH447X2103C can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15147